CLINICAL TRIAL: NCT02497781
Title: A Single Blind, Randomised, Multi-centre, Active Controlled, Trial To Evaluate Safety, Tolerability, Pharmacokinetics And Efficacy Of Ceftazidime And Avibactam Compared With Cefepime In Children From 3 Months To Less Than 18 Years Of Age With Complicated Urinary Tract Infections (Cutis)
Brief Title: Evaluation of Safety, Pharmacokinetics and Efficacy of Ceftazidime and Avibactam (CAZ-AVI ) Compared With Cefepime in Children From 3 Months to Less Than 18 Years of Age With Complicated Urinary Tract Infections (cUTIs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4280C00016; C3591005 (Other: Alias Study Number); 2014-003244-13 (EudraCT Number)
Record Dates: First submitted 2015-06-16; First posted 2015-07-15 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Complicated Urinary Tract Infections
Keywords: Complicated urinary tract infections (cUTIs)
MeSH Terms: interventions — avibactam, ceftazidime drug combination; Cefepime

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ceftazidime-avibactam (CAZ-AVI) (Experimental): CAZ-AVI to be administered every 8 hours as a 2-hour infusion (CAZ-AVI dose and frequency of IV administration will depend upon body weight and renal function)
  Interventions: Drug: Ceftazidime -avibactam
- Cefepime (Active Comparator): Patients randomised to receive cefepime should receive the dose, schedule and infusion duration as recommended in the local prescribing information or as prescribed by the investigator. The maximum dose of cefepime in any single infusion should not exceed 2000 mg
  Interventions: Drug: Cefepime

INTERVENTIONS:
Drug: Ceftazidime -avibactam — Patients randomised (3:1) to the CAZ-AVI or cefepime treatment
  Arms: ceftazidime-avibactam (CAZ-AVI)
Drug: Cefepime — Patients randomised (3:1) to the CAZ-AVI or cefepime treatment
  Arms: Cefepime

SUMMARY:
This study will assess the safety, tolerability and efficacy of ceftazidime and avibactam (CAZ-AVI )versus cefepime in children from 3 months to less than 18 years old with complicated urinary tract infections.

DETAILED DESCRIPTION:
This study will be a single-blind, randomised, multi-centre, active controlled trial. Patients aged from 3 months to less than 18 years with complicated urinary tract infections (cUTIs) will be randomised to 1 of 2 treatment groups (3:1 ratio): Ceftazidime and avibactam (CAZ AVI )or cefepime. Randomisation will be stratified by age cohort.

Patients will receive intravenous (IV) treatment for a minimum of 72 hours (3 full days, ie, 9 doses if given 3 times daily, or 6 doses if given twice daily) before having the option to switch to an oral therapy . The decision to switch to oral therapy is entirely at the Investigator's discretion, if the patient has good or sufficient clinical response, and the patient is tolerating oral fluids or food.

Patients will be assessed for safety and efficacy throughout the study, and blood samples will be taken for pharmacokinetic assessment. The duration of each patient's participation in the study will be a minimum of 27 days to a maximum of 50 days after start of study treatment including (intravenous treatment or oral switch therapy) 7 to 14 days of active treatment. The late follow-up visit (LFU) is to be performed 20 to 36 days after the last dose of any treatment.

The assessments at the test of cure (TOC) visit should be performed in person 8 to 15 days after last dose of any study drug Maximum duration of study drug or oral switch therapy is up to Day 14.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥3 calendar months to <18 years of age. Patients aged ≥3 calendar months to <1 year must have been born at term (defined as gestational age ≥37 weeks).
2. Written informed consent from parent(s) or other legally acceptable representative(s), and informed assent from patient (if age appropriate according to local regulations)
3. If female and has reached menarche, or has reached Tanner stage 3 development (even if not having reached menarche) (refer to Appendix E for further details on Tanner staging), the patient is authorised to participate in this clinical study if the following criteria are met:

   At screening:

   (i) (a) Patient reports sexual abstinence for the prior 3 months or reports use of at least 1 of the acceptable methods of contraception, including an intrauterine device (with copper banded coil), levonorgestrel intrauterine system (eg, Mirena®), or regular medroxyprogesterone injections (Depo-Provera®); or (b) Patient agrees to initiate sexual abstinence from the time of screening until 7 days after end of treatment with study drug; and (ii) Patient is advised to avoid conception from the time of screening until 7 days after receipt of study drug and agrees not to attempt pregnancy from the time of screening until 7 days after end of treatment with study drug; and (iii) Patient is provided guidelines regarding continuation of abstinence, initiation of abstinence, or about allowed contraception; and (iv) Patient has a negative serum β-human chorionic gonadotropin (β-hCG) test just prior to study entry. Since serum tests may miss an early pregnancy, relevant menstrual history and sexual history, including methods of contraception, should be considered. Note: if the result of the serum β-hCG test cannot be obtained prior to dosing of investigational product, a patient may be enrolled on the basis of a negative urine pregnancy test, though a serum β-hCG test result must still be obtained.
4. Patient has a clinically suspected and/or bacteriologically documented cUTI or acute pyelonephritis judged by the Investigator to be serious and requires the patient to be hospitalised for treatment with intravenous (IV) therapy
5. Patient has pyuria:

   Cohorts 1 to 3 as determined by a midstream clean catch or clean urethral catheterisation urine specimen with ≥10 white blood cells (WBCs) per high power field on standard examination of urine sediment or ≥10 WBCs/mm3 in unspun urine Cohort 4a and 4b as determined by a midstream clean catch or clean urethral catheterisation urine specimen or urine specimen obtained using urine collection pads(or supra-pubic collection if standard procedure in the assigned sites) ≥5 WBCs per high-power field on standard examination of urine sediment or ≥5 WBCs/mm3 in unspun urine
6. Patient has a positive urine culture: 1 midstream clean catch or clean urethral catheterisation urine specimen taken within 48 hours of randomisation containing ≥105 colony-forming units (CFU)/mL of a recognised uropathogen known to be susceptible to the IV study therapy (CAZ-AVI and cefepime) Note: If patients meet all of entry criteria except for positive urine culture as outlined above, the patients may be enrolled before urine culture results are available if the results are likely (based on urinalysis and clinical findings) to be positive and study drugs are considered appropriate empiric therapy. If a patient urine culture is negative after 24 or 48 hours of treatment but the patient is improving, the Investigator can keep the patient on treatment. If the urine culture is negative and the patient is not improving, study treatment will be stopped, and the patient will be followed for the rest of the study including undergoing all safety assessments until late follow up (LFU).
7. Demonstrates either acute pyelonephritis or complicated lower UTI as defined by the following criteria:

   1. Qualifying criteria: patients must have at least 1 of the following signs/symptoms (signs/symptoms must have onset or have worsened within 7 days of enrolment) in addition to pyuria:

      Dysuria (including perceived dysuria as referred by parent/caregiver) Urgency Frequency Abdominal pain Fever defined as oral temperature >38.5°C (or equivalent by other methods) with or without patient symptoms of rigor, chills, warmth Nausea Vomiting Irritability Loss of appetite Flank pain
   2. Or patients considered to have complicated UTI as indicated by 2 of the previous qualifying signs/symptoms in (a) plus at least 1 complicating factor from the following:

Recurrent UTI (2 or more within 12 months period) Obstructive uropathy that is scheduled to be surgically relieved during IV study therapy and before the EOT Functional or anatomical abnormality of the urogenital tract, including anatomic malformations or neurogenic bladder Vesicoureteral reflux Use of intermittent bladder catheterisation or presence of an indwelling bladder catheter for >48 hours prior to the diagnosis of cUTI Urogenital procedure (eg, cystoscopy or urogenital surgery) within the 7 days prior to study entry

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment or randomisation in the present study
3. Participation in another clinical study with an investigational product (IP) during the last 30 days before the first dose of IV study drug or have previously participated in the current study or in another study of CAZ-AVI (in which an active agent was received)
4. History of hypersensitivity reactions to carbapenems, cephalosporins, penicillins or other β-lactam antibiotics
5. Concurrent infection, including, but not limited to, central nervous system infection requiring systemic antibiotics in addition to the IV study drug therapy at the time of randomisation
6. Receipt of more than 24 hours of any systemic antibiotics after culture and before study drug therapy
7. Receipt of systemic antibiotics within 24 hours before obtaining the study qualifying pre-treatment baseline urine sample and before study drug therapy
8. The child is suspected or documented to have an infection caused by organisms resistant to the prophylactic antibiotics
9. A permanent indwelling bladder catheter or instrumentation including nephrostomy or current urinary catheter that will not be removed or anticipation of urinary catheter placement that will not be removed during the course of IV study drug therapy administration
10. Patient has suspected or known complete obstruction of any portion of the urinary tract, perinephric abscess, or ileal loops
11. Patient has had trauma to the pelvis or urinary tract
12. Patient has undergone renal transplantation
13. Patient has a condition or history of any illness that, in the opinion of the Investigator, would make the patient unsuitable for the study (eg, may confound the results of the study or pose additional risk in administering the study therapy to the patient)
14. Patient is considered unlikely to survive the 6 to 8 week study period or have a rapidly progressive illness, including septic shock that is associated with a high risk of mortality
15. At the time of randomisation, patient is known to have a cUTI caused by pathogens resistant to the antimicrobials planned to be used in the study
16. Presence of any of the following clinically significant laboratory abnormalities:

    1. Haematocrit <25% or haemoglobin <8 g/dL (<80 g/L, <4.9 mmol/L)
    2. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3×the age-specific upper limit of normal (ULN), or total bilirubin >2×ULN (except known Gilbert's disease) For a) to b): unless if these values are acute and directly related to the infectious process being treated.
17. Creatinine clearance <30 mL/min/1.73 m2 calculated using the child's measured height (length) and serum creatinine within the updated "bedside" Schwartz formula (Schwartz et al 2009):

    CrCl (mL/min/1.73m2)=0.413×height (length) (cm)/serum creatinine (mg/dL)
18. History of seizures, excluding well-documented febrile seizure of childhood
19. If female, currently pregnant or breast feeding

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (3):
  - Rady Children's Hospital San Diego, San Diego, California
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - ProMedica Toledo Children's Hospital, Toledo, Ohio
- Czechia (6):
  - Lekarna Oblastni nemocnice Kolin, a.s., Kolin III
  - Oblastni nemocnice Kolin, a.s., nemocnice Stredoceskeho kraje - Detske oddeleni, Kolin III
  - Krajska Zdravotni, A.S. - Nemocnice Most, O.Z., Detske A Dorostove Oddeleni, Most
  - Lekarna Nemocnice Most., O.Z., Most
  - Fakultni Nemocnice Ostrava - Klinika Detskeho Lekarstvi, Ostrava - Poruba
  - Lekarna Fakultni Nemocnice Ostrava, Ostrava - Poruba
- Greece (4):
  - General Children's Hospital "Agia Sofia", Goudi, Attica
  - General Children's Hospital of Athens "P. & A. Kyriakou", Goudi, Attica
  - "Hippokratio" General Hospital of Thessaloniki, Thessaloniki, Makedonia
  - University General Hospital of Larissa, Larissa, Thessaly
- Hungary (4):
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz - Rendelointezet, Gyermekinfektologiai Osztaly, Budapest
  - Toldy Ferenc Korhaz es Rendelointezet, Csecsemo- es Gyermekgyogyaszati Osztaly, Cegléd
  - Kanizsai Dorottya Korhaz, Csecsemo es Gyermekgyogyaszati Osztaly, Nagykanizsa
  - Tolna Megyei Balassa Janos Korhaz, Gyermekosztaly, Szekszárd
- Poland (2):
  - Uniwersytecki Dzieciecy Szpital Kliniczny im. L. Zamenhofa w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Wojewodzki Specjalistyczny Szpital im. dr W1. Bieganskiego, Lodz, Łódź Voivodeship
- Spitalul Clinic de Boli Infectioase si Tropicale "Dr. Victor Babes", Sectia B2 Boli Infectioase, Bucharest, Romania
- Russia (2):
  - State Autonomous Healthcare Institution of Kemerovo Region "Kemerovo Regional Clinical Hospital", Kemerovo
  - Federal State Budgetary Institution, Moscow
- Taiwan (4):
  - Hualien Tzu Chi Hospital Buddhist Tzu Chi Medical Foundation, Hualien City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- Turkey (Türkiye) (2):
  - Ege Universitesi Tip Fakultesi, Izmir
  - Celal Bayar Universitesi Hafsa Sultan Hastanesi, Manisa

REFERENCES:
- [Derived] Franzese RC, McFadyen L, Watson KJ, Riccobene T, Carrothers TJ, Vourvahis M, Chan PLS, Raber S, Bradley JS, Lovern M. Population Pharmacokinetic Modeling and Probability of Pharmacodynamic Target Attainment for Ceftazidime-Avibactam in Pediatric Patients Aged 3 Months and Older. Clin Pharmacol Ther. 2022 Mar;111(3):635-645. doi: 10.1002/cpt.2460. Epub 2021 Nov 22. PMID 34687548
- [Derived] Bradley JS, Roilides E, Broadhurst H, Cheng K, Huang LM, MasCasullo V, Newell P, Stone GG, Tawadrous M, Wajsbrot D, Yates K, Gardner A. Safety and Efficacy of Ceftazidime-Avibactam in the Treatment of Children >/=3 Months to <18 Years With Complicated Urinary Tract Infection: Results from a Phase 2 Randomized, Controlled Trial. Pediatr Infect Dis J. 2019 Sep;38(9):920-928. doi: 10.1097/INF.0000000000002395. PMID 31335570

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftazidime- Avibactam (CAZ-AVI): Participants with Creatinine clearance(CrCL) >=50 milliliter per minute (mL/min) received single IV infusion of CAZ/AVI for 2 hour in following manner: 1) Age 6 to less than (<)18 years: 2000 mg CAZ/500 mg AVI (body weight >=40 kg), 50 mg/kg CAZ/12.5 mg/kg AVI (body weight <40 kg), 2) Age 6 months to <6 years: 50 mg/kg CAZ/12.5 mg/kg AVI, 3) Age 3 months to <6 months: 40 mg/kg CAZ/10 mg/kg AVI. The infusion was administered to participants every 8 hours for a minimum of 72 hours and up to a maximum duration of 14 days. Dose of CAZ-AVI was reduced to 50 percent if CrCl of participant drops below to 50mL/min, and participant was removed from study therapy, if CrCl drops below 30mL/min. After having 72 hours of IV treatment, participants had option to switch to an oral therapy at investigator's discretion.
- Cefepime: Participants received intravenous (IV) infusion of cefepime, at a dose and frequency prescribed by investigator's (maximum dose of cefepime in any single infusion not exceed 2000 mg every 12 hours). After having 72 hours of IV treatment, participants had option to switch to an oral therapy at investigator's discretion.
Period: Overall Study
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Started | 68 | 29
Treated | 67 | 28
Completed | 64 | 26
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Randomised but not treated | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received any amount of IV study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime | Total
Number analyzed (Participants) | 67 | 28 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.08 (5.647) | 6.19 (6.072) | 6.12 (5.743)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 21 | 77
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 66 | 28 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 5 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 49 | 23 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Height [Mean (Standard Deviation); unit: centimeters] | 108.7 (34.40) | 108.9 (37.16) | 108.7 (35.03)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events between first dose of study drug and up to late follow-up (LFU) visit (20 to 36 days after last dose of study treatment [IV or oral]) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAE and non-SAE.
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Population: Safety analysis set included all randomized participants who received any amount of IV study medication (CAZ-AVI or Cefepime).
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
percentage of participants
  AEs | 53.7 | 53.6
  SAEs | 11.9 | 7.1

2. Primary Outcome: Percentage of Participants With Cephalosporin Class Effects and Additional Adverse Events (AEs)
Description: Percentage of participants with Cephalosporin class effects (defined as adverse event of special interest (AEoSI) within the safety topics (ST) of hypersensitivity/anaphylaxis) and additional AEs (which included AEs of diarrhea, renal disorder, hematological disorder and liver disorder relevant to the cephalosporin class within the safety topics (ST) based on MedDRA 20.0) were reported in this outcome measure.
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
percentage of participants
  AE in the ST of Diarrhea | 7.5 | 10.7
  AE in the ST of Hematological Disorders | 0 | 0
  AEoSI in the ST of Hypersensitivity/Anaphylaxis | 7.5 | 7.1
  AE in the ST of Liver Disorder | 1.5 | 0
  AE in the ST of Renal Disorder | 0 | 0

3. Primary Outcome: Change From Baseline in Pulse Rate at End of Intravenous Treatment (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 to 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
beats per minute
  Baseline | 111.5 (23.97) | 119.1 (27.08)
  Change at EOIV | -11.9 (18.65) | -17.1 (24.58)

4. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at End of Intravenous Treatment (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 to 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
millimeter of mercury (mmHg)
  SBP: Baseline | 105.6 (14.88) | 111.9 (14.61)
  SBP: Change at EOIV | -1.0 (15.11) | -5.4 (14.53)
  DBP: Baseline | 62.6 (12.68) | 69.1 (9.28)
  DBP: Change at EOIV | 0.9 (15.41) | -5.0 (7.50)

5. Primary Outcome: Change From Baseline in Respiratory Rate at End of Intravenous Treatment (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 to 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
breaths per minute
  Baseline | 25.8 (5.96) | 27.0 (8.46)
  Change at EOIV: number analyzed (Participants) | 67 | 27
  Change at EOIV | -2.5 (4.64) | -2.6 (7.96)

6. Primary Outcome: Change From Baseline in Body Temperature at End of Intravenous Treatment (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 to 15)
Population: Safety analysis set included all randomized participants who received any amount of IV study medication (CAZ-AVI or Cefepime). Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 66 | 28
degree Celsius
  Baseline | 37.67 (1.043) | 37.49 (1.031)
  Change at EOIV | -1.15 (1.096) | -0.90 (1.036)

7. Primary Outcome: Percentage of Participants With Abnormal Physical Examination Findings at End of Intravenous Treatment (EOIV) Visit
Description: Physical examination included an assessment of the following: general appearance, skin, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, respiratory system, cardiovascular system, abdomen, musculoskeletal system (including spine and extremities), and neurological system. Participants with new or aggravated abnormal physical examination findings with regard to baseline findings were reported. Abnormality in physical examinations were based on blinded observer's discretion. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: EOIV visit (anytime from Day 4 to 15)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
percentage of participants
  Abdomen | 0 | 3.6
  Cardiovascular System | 1.5 | 0
  General Appearance | 0 | 0
  Head and Neck | 1.5 | 3.6
  Lymph Nodes | 0 | 3.6
  Musculoskeletal System | 0 | 0
  Neurological System | 0 | 0
  Respiratory System | 3.0 | 0
  Skin | 3.0 | 7.1
  Thyroid | 0 | 0

8. Primary Outcome: Change From Baseline in Body Weight at End of Intravenous Treatment (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 to 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
kilogram
  Baseline | 24.55 (19.361) | 25.24 (21.527)
  Change at EOIV: number analyzed (Participants) | 66 | 28
  Change at EOIV | -0.08 (0.613) | 0.14 (0.510)

9. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Abnormalities in Laboratory Parameters
Description: Criteria for potentially clinically significant laboratory abnormalities: hematology (platelets: <0.4*lower limit of normal [LLN], >2*upper limit of normal [ULN], >40% decrease from baseline [DFB],>100% Increase from baseline [IFB]; Chemistry (Bicarbonate: <0.7*LLN, >1.3*ULN, >50% DFB, >30% IFB).
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 62 | 26
percentage of participants
  Chemistry: Bicarbonate: number analyzed (Participants) | 51 | 23
  Chemistry: Bicarbonate | 2.0 | 0
  Hematology: Platelets | 1.6 | 0

10. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Abnormalities in Electrocardiogram (ECG) Parameters
Description: PCS criteria for abnormal value of ECG parameters: QT interval >=450 milliseconds (msec); 480 msec; >=500 msec; Increase from baseline (IFB) of >=30 msec; >=60 msec and >90 msec; Decrease from baseline (DFB) of >=30 msec; >=60 msec and >90 msec. QT interval using Bazett's correction (QTcB): >=450 milliseconds (msec); 480 msec; >=500 msec; Increase from baseline (IFB) of >=30 msec; >=60 msec and >90 msec; DFB of >=30 msec; >=60 msec and >90 msec. QT interval using Fridericia's correction (QTcF): >=450 msec; 480 msec; >=500 msec; IFB of >=30 msec; >=60 msec and >90 msec; DFB of >=30 msec; >=60 msec and >90 msec. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline until the EOIV visit (anytime from Day 4 to 15)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
percentage of participants
  QT Interval : >450 msec | 0 | 0
  QT Interval : >480 msec | 0 | 0
  QT Interval : >500 msec | 0 | 0
  Maximum IFB QT Interval : > 30 msec | 19.4 | 14.3
  Maximum IFB QT Interval : > 60 msec | 7.5 | 3.6
  Maximum IFB QT Interval : >90 msec | 3.0 | 0
  Maximum DFB QT Interval : > 30 msec | 9.0 | 17.9
  Maximum DFB QT Interval : > 60 msec | 4.5 | 0
  Maximum DFB QT Interval : > 90 msec | 1.5 | 0
  QTcB Interval : >450 msec | 16.4 | 3.6
  QTcB Interval : >480 msec | 11.9 | 0
  QTcB Interval : >500 msec | 7.5 | 0
  Maximum IFB QTcB Interval : > 30 msec | 17.9 | 14.3
  Maximum IFB QTcB Interval : > 60 msec | 7.5 | 3.6
  Maximum IFB QTcB Interval : > 90 msec | 3.0 | 0
  Maximum DFB QTcB Interval : > 30 msec | 10.4 | 7.1
  Maximum DFB QTcB Interval : > 60 msec | 6.0 | 3.6
  Maximum DFB QTcB Interval : > 90 msec | 1.5 | 3.6
  QTcF Interval : >450 msec | 6.0 | 0
  QTcF Interval : >480 msec | 6.0 | 0
  QTcF Interval : >500 msec | 6.0 | 0
  Maximum IFB QTcF Interval : > 30 msec | 17.9 | 14.3
  Maximum IFB QTcF Interval : > 60 msec | 3.0 | 3.6
  Maximum IFB QTcF Interval : > 90 msec | 3.0 | 0
  Maximum DFB QTcF Interval : > 30 msec | 9.0 | 10.7
  Maximum DFB QTcF Interval : > 60 msec | 3.0 | 3.6
  Maximum DFB QTcF Interval : > 90 msec | 1.5 | 0

11. Primary Outcome: Percentage of Participants With Creatinine Clearance (CrCl) at Day 7
Description: CrCl is a measure of glomerular filtration rate (GMFR), an index of kidney function. It is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Percentage of participants with CrCl in the following categories were reported: <30 mL/min/1.73 m^2, >=30 to <50 mL/min/1.73 m^2, >=50 mL/min/1.73 m^2 to <80 mL/min/1.73 m^2, and >=80 mL/min/1.73 m^2.
Time Frame: Day 7
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
percentage of participants
  CrCl: <30mL/min/1.73 m^2 | 0 | 0
  CrCl: >=30 to <50mL/min/1.73 m^2 | 0 | 0
  CrCl: >=50 to <80mL/min/1.73 m^2 | 11.1 | 0
  CrCl: >=80mL/min/1.73 m^2 | 88.9 | 100

12. Primary Outcome: Percentage of Participants With Creatinine Clearance (CrCl) at End of Intravenous Treatment (EOIV) Visit
Description: CrCl is a measure of glomerular filtration rate (GMFR), an index of kidney function. It is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Percentage of participants with CrCl in the following categories were reported: <30 mL/min/1.73 m^2, >=30 to <50 mL/min/1.73 m^2, >=50 mL/min/1.73 m^2 to <80 mL/min/1.73 m^2, and >=80 mL/min/1.73 m^2. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: EOIV visit (anytime from Day 4 to 15)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
percentage of participants
  CrCl: <30mL/min/1.73 m^2 | 0 | 0
  CrCl: >=30 to <50mL/min/1.73 m^2 | 0 | 0
  CrCl: >=50 to <80mL/min/1.73 m^2 | 20.0 | 13.6
  CrCl: >=80mL/min/1.73 m^2 | 80.0 | 86.4

13. Primary Outcome: Percentage of Participants With Creatinine Clearance (CrCl) at Test of Cure (TOC) Visit
Description: CrCl is a measure of glomerular filtration rate (GMFR), an index of kidney function. It is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Percentage of participants with CrCl in the following categories were reported: <30 mL/min/1.73 m^2, >=30 to <50 mL/min/1.73 m^2, >=50 mL/min/1.73 m^2 to <80 mL/min/1.73 m^2, and >=80 mL/min/1.73 m^2. TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral).
Time Frame: TOC visit (up to a maximum study duration of 50 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 67 | 28
percentage of participants
  CrCl: <30mL/min/1.73 m^2 | 0 | 0
  CrCl: >=30 to <50mL/min/1.73 m^2 | 0 | 0
  CrCl: >=50 to <80mL/min/1.73 m^2 | 25.0 | 41.7
  CrCl: >=80mL/min/1.73 m^2 | 75.0 | 58.3

14. Secondary Outcome: Plasma Concentrations of Ceftazidime and Avibactam
Time Frame: 15, 30-90, 300-360 minutes post-dose on Day 3
Population: PK analysis set included all randomized participants who received any amount of CAZ-AVI and had at least 1 CAZ and/ or AVI plasma measurement available. This outcome measure was not planned to be analyzed for Cefepime receiving cohort, as pre-specified in protocol.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI)
Number analyzed (Participants) | 64
nanogram per milliliter
  Ceftazidime: 15 minute post-dose on Day 3: number analyzed (Participants) | 62
  Ceftazidime: 15 minute post-dose on Day 3 | 61411.2 (39276.40)
  Ceftazidime: 30-90 minute post-dose on Day 3: number analyzed (Participants) | 59
  Ceftazidime: 30-90 minute post-dose on Day 3 | 47638.5 (31948.31)
  Ceftazidime:300-360minute post-dose on Day 3: number analyzed (Participants) | 62
  Ceftazidime:300-360minute post-dose on Day 3 | 7285.7 (11396.88)
  Avibactam: 15 minute post-dose on Day 3: number analyzed (Participants) | 62
  Avibactam: 15 minute post-dose on Day 3 | 9577.4 (6922.76)
  Avibactam: 30-90 minute post-dose on Day 3: number analyzed (Participants) | 59
  Avibactam: 30-90 minute post-dose on Day 3 | 7046.4 (6060.75)
  Avibactam: 300-360 minute post-dose on Day 3: number analyzed (Participants) | 62
  Avibactam: 300-360 minute post-dose on Day 3 | 936.3 (1499.00)

15. Secondary Outcome: Percentage of Participants With Favourable Clinical Response (CR): Intent-to-treat (ITT) Analysis Population
Description: Favorable CR was defined as a CR of improvement and cure(at end of 72 hours(hr) and EOIV) and a CR of cure(at EOT and TOC).Cure is resolution of all acute signs/symptoms of cUTI/improvement to such an extent that no further antimicrobial therapy required.Improvement is:1)at end of 72hr study drug treatment: improvement but not enough to switch to oral therapy and still on IV study drug at end of 72hr and meet following criterion: Absence of new signs/symptoms, and improvement in at least 1 symptom/sign(ie, fever,pain,tenderness,elevated WBCs,elevated CRP) from Baseline,and with no worsening of any symptom/sign. 2) at EOIV: participants who switched to oral therapy and had afebrile(temperature<=38.0°C) for >=24hr;absence of new and improvement in at least 1 symptom/sign from Baseline and worsening of none.EOT visit occurred within 48hr after completion of the last dose of oral switch therapy or at time of premature discontinuation/early withdrawal from study(if on oral switch therapy).
Time Frame: End of 72 hours study drug treatment, EOIV visit (anytime from Day 4 to 15), EOT visit (up to Day 16), TOC visit (up to a maximum study duration of 50 days)
Population: ITT analysis population included all participants who had been assigned a randomized treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 68 | 29
percentage of participants
  End of 72 hours | 88.2 [79.0 to 94.3] | 86.2 [70.5 to 95.2]
  EOIV | 91.2 [82.7 to 96.2] | 89.7 [74.9 to 97.0]
  EOT | 88.2 [79.0 to 94.3] | 89.7 [74.9 to 97.0]
  TOC | 86.8 [77.2 to 93.2] | 82.8 [66.3 to 93.1]

16. Secondary Outcome: Percentage of Participants With Favourable Clinical Response (CR): Microbiological ITT (Micro-ITT) Analysis Population
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Micro-ITT analysis population included all randomized participants who had at least 1 gram negative typical pathogen (in the urine) at baseline known to cause cUTI and no gram positive pathogen (in the urine) at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 54 | 23
percentage of participants
  End of 72 hours | 90.7 [80.9 to 96.4] | 95.7 [81.4 to 99.5]
  EOIV | 96.3 [88.6 to 99.2] | 95.7 [81.4 to 99.5]
  EOT | 90.7 [80.9 to 96.4] | 95.7 [81.4 to 99.5]
  TOC | 88.9 [78.5 to 95.2] | 82.6 [63.8 to 93.8]

17. Secondary Outcome: Percentage of Participants With Favourable Clinical Response (CR) at End of 72 Hours Treatment: Clinically Evaluable (CE) Analysis Set at 72 Hours
Description: Favourable clinical response was defined as a CR of improvement and cure. Cure was defined as resolution of all acute signs and symptoms of complicated urinary tract infections (cUTIs) or improvement to such an extent that no further antimicrobial therapy was required. Clinical Improvement included all the participants who had improvement but not enough to switch to oral therapy and were still on IV study drug at End of 72 hours and had meet the following criterion: absence of new signs and symptoms, and improvement in at least 1 symptom or sign (fever, pain, tenderness, elevated WBCs, elevated CRP) from baseline, and with no worsening of any symptom or sign.
Time Frame: End of 72 hours study drug treatment on Day 1
Population: CE analysis set at 72hr: participants who had at least 1 gram negative typical pathogen (in urine) at baseline known to cause cUTI, no gram positive pathogen (in urine) at baseline, confirmed diagnosis of cUTI, >=48hr of IV study drug, unless discontinued due to treatment-limiting AE, no important protocol deviations and no concomitant antibiotics.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 47 | 21
percentage of participants | 100 [94.8 to 100] | 95.2 [79.8 to 99.5]

18. Secondary Outcome: Percentage of Participants With Favourable Clinical Response (CR) at End of Intravenous Treatment (EOIV) Visit: Clinically Evaluable (CE) Analysis Set at EOIV
Description: Favourable clinical response was defined as a CR of improvement and cure. Cure was defined as resolution of all acute signs and symptoms of complicated urinary tract infections (cUTIs) or improvement to such an extent that no further antimicrobial therapy was required. Clinical Improvement included all the participants who had switched to oral therapy and had meet the following criterion: afebrile (temperature <=38.0°C) for at least 24 hours, absence of new and improvement in at least 1 symptom or sign (fever, pain, tenderness, elevated WBCs, elevated c-reactive-protein) from baseline and worsening of none. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: EOIV visit (anytime from Day 4 to 15)
Population: CE analysis set at EOIV: participants >=1 gram negative typical pathogen known to cause cUTI, no gram positive pathogen (in urine) at baseline, confirmed cUTI diagnosis, >=48 h of IV study drug, unless discontinued due to AE, no important protocol deviations, no concomitant antibiotic, had clinical response of cure, improvement or failure at EOIV.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 52 | 22
percentage of participants | 98.1 [91.4 to 99.8] | 95.5 [80.7 to 99.5]

19. Secondary Outcome: Percentage of Participants With Favourable Clinical Response (CR) at End of Treatment (EOT) Visit: Clinically Evaluable (CE) Analysis Set at EOT
Description: Favourable clinical response was defined as a CR cure. Cure was defined as resolution of all acute signs and symptoms of complicated urinary tract infections (cUTIs) or improvement to such an extent that no further antimicrobial therapy was required. EOT visit occurred within 48hr after completion of the last dose of oral switch therapy or at time of premature discontinuation/early withdrawal from study(if on oral switch therapy).
Time Frame: EOT visit (up to Day 16)
Population: CE analysis set at EOT: participants >=1 gram negative typical pathogen known to cause cUTI, no gram positive pathogen (in urine) at baseline, confirmed cUTI diagnosis, >=48hr of IV study drug, unless discontinued due to AE, no important protocol deviations, no concomitant antibiotic, had clinical response of cure, improvement or failure at EOT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 49 | 19
percentage of participants | 98.0 [90.9 to 99.8] | 94.7 [77.9 to 99.4]

20. Secondary Outcome: Percentage of Participants With Favourable Clinical Response (CR) at TOC: Clinically Evaluable (CE) Analysis Set at TOC
Description: Favourable clinical response was defined as resolution of all acute signs/symptoms of cUTIs or improvement to such an extent that no further antimicrobial therapy was needed. Participants who met the following criterion: Incomplete resolution or worsening of cUTI signs or symptoms or development of new signs or symptoms requiring alternative non-study antimicrobial therapy or death in which cUTI was contributory. TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral).
Time Frame: TOC visit (up to a maximum study duration of 50 days)
Population: CE analysis set at TOC: participants >=1 gram negative typical pathogen known to cause cUTI, no gram positive pathogen (in urine) at baseline, confirmed cUTI diagnosis, >=48hr of IV study drug, unless discontinued due to AE, no important protocol deviations, no concomitant antibiotic, had clinical response of cure, improvement or failure at TOC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 49 | 20
percentage of participants | 93.9 [84.6 to 98.2] | 85.0 [65.1 to 95.6]

21. Secondary Outcome: Percentage of Participants With Favourable Clinical Response (CR): Microbiologically Evaluable (ME) Analysis Population
Description: as for outcome 15
Time Frame: EOIV visit (anytime from Day 4 to 15), EOT visit (up to Day 16), TOC visit (up to a maximum study duration of 50 days)
Population: ME analysis set: participants >=1gram(-ve) and no gram(+ve) pathogen (in urine) at baseline, confirmed cUTI diagnosis, had >=48hr IV study drug, unless discontinued due to AE, no important protocol deviation, concomitant antibiotic, >=1gram(-ve) typical UTI bacterial pathogen at Baseline susceptible to study drug and MR which was not indeterminate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 41 | 16
percentage of participants
  EOIV: number analyzed (Participants) | 35 | 16
  EOIV | 100 [93.1 to 100] | 100 [85.7 to 100]
  EOT: number analyzed (Participants) | 39 | 14
  EOT | 100 [93.8 to 100] | 100 [83.8 to 100]
  TOC | 92.7 [81.7 to 97.9] | 87.5 [65.6 to 97.3]

22. Secondary Outcome: Percentage of Participants With Favourable Microbiological Response: Microbiological Intent-to-treat (Micro-ITT) Population
Description: Favourable microbiological response was achieved when all baseline pathogens were eradicated. EOIV visit occurred within 24 hours after completion of last infusion of the study drug. EOT visit occurred within 48 hours after completion of the last dose of oral switch therapy or at time of premature discontinuation/early withdrawal from study if on oral switch therapy (which occurred within the maximum study treatment duration of 14 days).
Time Frame: EOIV visit (Day 4 to 15), EOT visit(up to Day 16)
Population: Micro-ITT analysis population included all randomized participants who had at least 1 gram negative typical pathogen (in the urine) at baseline known to cause cUTI and no gram cUTI and no gram positive pathogen (in the urine) at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 54 | 23
percentage of participants
  EOIV | 81.5 | 78.3
  EOT | 83.3 | 73.9

23. Secondary Outcome: Percentage of Participants With Favourable Microbiological Response: Microbiologically Evaluable (ME) Analysis Population
Description: as for outcome 22
Time Frame: EOIV visit (Day 4 to 15), EOT visit (up to Day 16)
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 39 | 16
percentage of participants
  EOIV: number analyzed (Participants) | 35 | 16
  EOIV | 97.1 | 100
  EOT: number analyzed (Participants) | 39 | 14
  EOT | 97.4 | 100

24. Secondary Outcome: Percentage of Participants With Clinical Relapse at Late Follow-up (LFU) Visit: Clinically Evaluable (CE) Analysis Set at LFU
Description: A participant was said to have clinical relapse if met either 1 of the following criteria: reappearance or worsening of signs and symptoms of cUTI that required further antimicrobial therapy and/or surgery or death after TOC in which cUTI was contributory. LFU visit occurred within 20 to 36 days after last dose of study treatment (IV or oral).
Time Frame: LFU visit (anytime up to a maximum study duration of 50 days)
Population: CE analysis set at LFU: participants >=1gram negative typical pathogen known to cause cUTI, no gram positive pathogen (in urine) at baseline, confirmed cUTI diagnosis, >=48hr of IV study drug, unless discontinued due to AE, no important protocol deviations, no concomitant antibiotic,were evaluated for clinical response of sustained cure or relapse.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 52 | 22
percentage of participants | 6.8 | 0

25. Secondary Outcome: Percentage of Participants With Clinical Relapse at Late Follow-up (LFU) Visit: Microbiologically Evaluable (ME) Analysis Set at LFU
Description: A participant was said to have clinical relapse if met either 1 of the following criteria: reappearance or worsening of signs and symptoms of cUTI that required further antimicrobial therapy and/or surgery, or death after TOC in which cUTI was contributory. LFU visit occurred within 20 to 36 days after last dose of study treatment (IV or oral).
Time Frame: LFU visit (anytime up to a maximum study duration of 50 days)
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 16 | 9
percentage of participants | 12.5 | 0

26. Secondary Outcome: Percentage of Participants With Emergent Infections: Microbiological Intent-to-treat (Micro-ITT) Population
Description: Emergent infections were categorized as super-infection and new infections. Superinfection: A urine culture identified pathogen other than a baseline pathogen during the course of active treatment with study therapy along with worsening signs and symptoms of infection requiring alternative antimicrobial therapy. New infection: A urine culture identified pathogen other than a baseline pathogen at any time after study treatment had finished along with worsening signs and symptoms of infection requiring alternative antimicrobial therapy. Percentage of participants with any (super infections or new infections) of the infections were reported.
Time Frame: Baseline up to 50 days
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 54 | 23
percentage of participants | 5.6 | 0

27. Secondary Outcome: Percentage of Participants With Emergent Infections: Microbiologically Evaluable (ME) Analysis Population
Description: as for outcome 26
Time Frame: Baseline up to 50 days
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 41 | 16
percentage of participants | 7.3 | 0

28. Secondary Outcome: Percentage of Participants With Favourable Combined Response: Microbiological Intent-to-treat (Micro-ITT) Population
Description: Combined response was the combined assessment of clinical response and microbiological response. Favorable clinical response was defined as a clinical response of improvement and cure (at EOIV) and a clinical response of cure (at TOC). Cure defined as: resolution of all acute signs/symptoms of cUTI/improvement to such an extent that no further antimicrobial therapy required. Improvement defined as: participants who switched to oral therapy and had afebrile (temperature<=38.0°C) for >=24 hr; absence of new and improvement in at least 1 symptom or sign (ie, fever, pain, tenderness, elevated WBCs, elevated CRP) from Baseline and worsening of none. Favourable microbiological response was absence of the original baseline pathogen in source specimen. EOIV visit occurred within 24 hours after completion of last infusion of the study drug. TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral).
Time Frame: EOIV visit (Day 4 to 15), TOC visit (up to a maximum study duration of 50 days)
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 54 | 23
percentage of participants
  Favourable at EOIV | 79.6 | 78.3
  Favourable at TOC | 72.2 | 60.9

29. Secondary Outcome: Percentage of Participants With Combined Response: Microbiologically Evaluable (ME) Analysis Population
Description: as for outcome 28
Time Frame: EOIV visit (Day 4 to 15), TOC visit (up to a maximum study duration of 50 days)
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
Number analyzed (Participants) | 41 | 16
percentage of participants
  Favourable at EOIV: number analyzed (Participants) | 35 | 16
  Favourable at EOIV | 97.1 | 100
  Favourable at TOC | 80.5 | 68.8

ADVERSE EVENTS:
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) | Cefepime
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/28
Serious Adverse Events (participants affected / at risk) | 8/67 | 2/28
Other Adverse Events (participants affected / at risk) | 13/67 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime- Avibactam (CAZ-AVI) (N=67) | Cefepime (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime- Avibactam (CAZ-AVI) (N=67) | Cefepime (N=28)
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Rhinitis (Infections and infestations) | 4 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT02497781/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT02497781/SAP_001.pdf